CLINICAL TRIAL: NCT00323076
Title: A Phase I/II Imaging Study of 1-a-D-(5-deoxy-5-[18]F-fluoroarabinofuranosyl)-2-nitroimidazole ([18]F-FAZA) in Patients With Known Squamous Cell Carcinoma of the Head & Neck, Small Cell and Non-Small Cell Carcinoma of the Lung, Lymphoma, Glioblastoma Multiforme, Neuroendocrine Tumours or Renal Cell Carcinoma
Brief Title: [18]F-FAZA PET Imaging Study in Patients With Cancer of the Head & Neck, Lung, Renal Cell, Brain, Lymphoma and Neuroendocrine Tumours
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Retirement of former Qualified Investigator and lack of resources to complete study.
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DX-FAZ-001
Record Dates: First submitted 2006-05-05; First posted 2006-05-09 (Estimated); Last update posted 2019-08-26 (Actual); Status verified 2019-02

CONDITIONS: Renal Cell Carcinoma; Neuroendocrine Tumours
MeSH Terms: conditions — Carcinoma, Renal Cell; Neuroendocrine Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): 18F-FAZA PET Imaging
  Interventions: Drug: 18F-FAZA PET Imaging

INTERVENTIONS:
Drug: 18F-FAZA PET Imaging — Phase I: 110-600 MBq per injection. A single injection of 18F-FAZA and PET scan will be permitted per patient.
  Phase II: 110-600 MBq per injection. Up to three separate injections of 18F-FAZA and PET scans will be permitted per patient.

SUMMARY:
Positron Emission Tomography (PET) is a Nuclear Medicine procedure that uses positron emitting radiolabeled tracer molecules to visualize biological activity. The presence of hypoxia (low oxygen) is associated with poor prognosis in a variety of tumour types and treatment strategies targeting hypoxic cells have been developed. The PET tracer [18]F-FAZA can identify hypoxic areas, and changes in uptake during treatment may predict tumour response.

DETAILED DESCRIPTION:
The proposed clinical trial will be a Phase I/II imaging, open label, single site study. In Phase I, one 18F-FAZA PET scan will be conducted in patients with known squamous cell carcinoma of the Head & Neck, SCLC, NSCLC, lymphoma, GGM, neuroendocrine tumours or renal cell carcinoma. In Phase II, three 18F-FAZA PET scans will be done on patients with the above tumours as follows: one pre-treatment, one mid course and one post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female greater than or equal to 16 years of age.
* If female of child-bearing potential and outside of the window of 10 days since the first day of the last menstrual period, a negative pregnancy test is required.
* Patients with known primary or suspected metastatic squamous cell carcinoma of the head and neck, non-small cell or small cell carcinoma of the lung, lymphoma, GBM (greater than or equal to 3 glioma), neuroendocrine tumours, or renal cell carcinoma with at least one lesion >1 cm in diameter.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2006-09-12 (Actual); Primary Completion 2019-02-04 (Actual); Study Completion 2019-02-04 (Actual)

PRIMARY OUTCOMES:
Phase I: demonstrate the safety of 18F-FAZA manufactured at the Edmonton Radiopharmaceutical Centre/Edmonton PET Centre. Phase II: determine the general biodistribution pattern of18F-FAZA. | Phase I: 2 years, Phase II: 5 years
  Phase I: Pre-injection and post-imaging vital signs, blood haematology and blood chemistry, adverse event collection.
  Phase II: The location and relative uptake of normal and abnormal 18F-FAZA biodistribution patterns will be determined.

SECONDARY OUTCOMES:
Determine the relative tumour uptake of 18F-FAZA | 5 years
  Measure relative uptake scores (RUS) and tumour to background ratios (T/B) and correlate this uptake to disease progression, disease-free survival, overall survival and response to treatment over 12 months of follow-up.
Confirm the safety of 18F-FAZA manufactured at the Edmonton Radiopharmaceutical Centre/Edmonton PET Centre | 5 years
  Adverse event collection

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel W Hudson, MD, Principal Investigator — Cross Cancer Institute
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada

REFERENCES:
- [Background] Postema EJ, McEwan AJ, Riauka TA, Kumar P, Richmond DA, Abrams DN, Wiebe LI. Initial results of hypoxia imaging using 1-alpha-D: -(5-deoxy-5-[18F]-fluoroarabinofuranosyl)-2-nitroimidazole ( 18F-FAZA). Eur J Nucl Med Mol Imaging. 2009 Oct;36(10):1565-73. doi: 10.1007/s00259-009-1154-5. Epub 2009 May 9. PMID 19430784